CLINICAL TRIAL: NCT00086528
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL647 Administered Orally to Subjects With Solid Tumors
Brief Title: Safety and Pharmacokinetics of XL647 Administered Orally to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL647-001
Record Dates: First submitted 2004-07-02; First posted 2004-07-07 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL647 — Administered orally as a solution with mass-based dosing in early cohorts or as 50-mg tablets at a fixed dose at the MTD. A minimum of 3 subjects was planned for each dosing cohort with dose escalation dependent on subject tolerance of the prior dose. During the Treatment Period, subjects in each cohort were administered a single dose of XL647 on Day 1 followed by a 72-hour period of observation. If there were no XL647-related dose limiting toxicities, subjects received 5 daily doses of XL647 on Days 4-8. Twenty-one days after the initial dose, in the absence of unacceptable toxicity or disease progression, subjects could enter a Treatment Extension Period that consisted of repeated 2-week cycles of five oral doses of XL647 followed by a 9-day observation period.
  Other Names: KD019

SUMMARY:
The primary objective of this study is as follows:

* To evaluate the safety and tolerability of XL647 administered orally as a single dose and as repeat doses in subjects with solid tumors.

The secondary objectives of this study are as follows:

* To evaluate the plasma pharmacokinetics of XL647 administered orally as a single dose and as repeat doses in subjects with solid tumors,
* To estimate renal elimination of XL647 administered orally as a single dose in subjects with solid tumors.

The exploratory objective of this study is as follows:

* To assess the pharmacodynamic effects of XL647 administration in plasma and peripheral blood cells.

In addition, subjects may be eligible to enter a Treatment Extension Period. The following information will be obtained from this part of the study:

* Long-term safety and tolerability of XL647 after repeat administration,
* Tumor response after repeat administration of XL647.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed malignancy that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective,
* The subject has disease that is assessable by tumor marker, physical, or radiologic means,
* The subject is ≥18 years old,
* There have been at least 4 weeks since prior chemotherapy or radiation therapy (6 weeks if the last treatment regimen included BCNU or mitomycin C),
* The subject has an ECOG performance status ≤2 (Karnofsky >60%),
* The subject has a life expectancy of ≥3 months,
* The subject has normal organ and marrow function (hemoglobin >10g/dL, leukocytes >3,000/mL, absolute neutrophil count >1,500/µL, platelets >100,000/µL, total bilirubin within normal institutional limits of normal,AST (SGOT)/ALT(SGPT) <2.5 times the upper limit of normal, and creatinine within normal limits,
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document,
* Sexually active subjects (both male and female) must use an accepted method of contraception during the course of the study,
* Female subjects of childbearing potential (pre-menopausal) must have a negative pregnancy test.

Exclusion Criteria:

* The subject has had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or has not recovered from AEs due to agents administered more than 4 weeks earlier,
* The subject has received another investigational agent within 30 days (or 5.5 half-lives) of the first dose of study drug,
* The subject has known brain metastases,
* The subject has a corrected QT interval (QTc) of >0.44 seconds,
* The subject has a history of allergic reactions attributed to aspartame or to any other component in the formulation vehicle,
* The subject has an uncontrolled intercurrent illness including,but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements,
* The subject is pregnant or nursing,
* The subject is known to be positive for the human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of XL647 administered orally as a single dose and as repeat doses | First treatment until 30 days post last treatment

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics of XL647 administered orally as a single dose and as repeat dose | At various time points between pre-treatment and post last treatment
To estimate renal elimination of XL647 administered orally as a single dose in subjects with solid tumors | At various time points between pre-treatment and post last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harold Keer, M.D., Ph.D., Study Director — Exelixis, Inc. (Study Sponsor)
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Das M, Padda SK, Frymoyer A, Molina J, Adjei A, Lensing JL, Miles D, Sikic BI, Wakelee HA. A safety, tolerability, and pharmacokinetic analysis of two phase I studies of multitargeted small molecule tyrosine kinase inhibitor XL647 with an intermittent and continuous dosing schedule in patients with advanced solid malignancies. Cancer Chemother Pharmacol. 2018 Sep;82(3):541-550. doi: 10.1007/s00280-018-3646-0. Epub 2018 Jul 20. PMID 30030583